CLINICAL TRIAL: NCT05839808
Title: Reliability and Validity of the Turkish Version of the Stroke Exercise Preference Inventory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 83116987-272
Record Dates: First submitted 2023-04-18; First posted 2023-05-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: Reliability; Validity; Stroke; Stroke Exercise Preference Inventory
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individuals who have had a stroke (Other): To evaluate the validity and reliability of the Stroke Exercise Preference Inventory
  Interventions: Other: Reliability and validity study

INTERVENTIONS:
Other: Reliability and validity study — To evaluate the validity and reliability of the Stroke Exercise Preference Inventory

SUMMARY:
With this study, it will be proven whether the Turkish version of the Stroke Exercise Preference Inventory is valid and reliable in evaluating the exercise preferences of individuals who have had a stroke.

DETAILED DESCRIPTION:
Version, validity, and reliability studies are frequently encountered in the literature. However, there is no scale that evaluates the exercise preferences of individuals who have had a stroke among the measurement tools whose Turkish version, validity, and reliability studies have been carried out. The Stroke Exercise Preference Inventory is an outcome scale for questioning exercise preferences in individuals who have had a stroke. It is functional for the development and planning of exercise programs for individuals who have had a stroke. This scale will both fill the gap in the Turkish literature in terms of the parameters it evaluates and will be the first in this context. In terms of its application, it is a useful inventory in this field. Considering the absence of a measurement tool developed in Turkish or adapted to Turkish for the assessment of exercise preferences of individuals with stroke, the aim of this study is to evaluate the validity and reliability of the Turkish version of the self-administered Stroke Exercise Preference Inventory, designed to question exercise preferences in Turkish individuals with stroke, to perform cross-cultural adaptation study, and to question the suitability of the Turkish version for Turkish society and the effectiveness of its clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Who have had a stroke,
* Good cognitive status,
* Can speak, read, write Turkish.

Exclusion Criteria:

* Pregnant,
* Who cannot speak, read or write Turkish.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Exercise preference | through study completion, an average of 6 month
  The Stroke Exercise Preference Inventory was developed in 2016 as an inventory consisting of 13 items. The inventory also includes 9 items that assess exercise barriers. The Stroke Exercise Preference Inventory is very useful and beneficial for clinicians in terms of determining the exercise preferences of individuals who have had a stroke and questioning the thoughts of the individual in continuing the exercise and rehabilitation program. It is functional for the development and planning of exercise programs for individuals who have had a stroke. Inventory scores as a percentage. And the decreasing score indicates the negativity of participation and view of the exercise.
Cognitive status | through study completion, an average of 6 month
  The Mini Mental Test will be used to quantitatively assess cognitive performance. It consists of eleven items gathered under five main headings as orientation, recording memory, attention and calculation, recall and language, and is evaluated out of a total score of 30. A minimum of 24 points must be obtained.
Functional ambulation | through study completion, an average of 6 month
  The Functional Ambulation Classification will be used for the evaluation of ambulation in individuals. The Functional Ambulation Classification shows the support surfaces that walking patients receive. It is valuable when starting to step and walk from the immobility period. It is calculated over a total of 6 categories by scoring between 0 and 5.
Activity status | through study completion, an average of 6 month
  The Frenchay Activities Index is a 15-item index that was created to collect information about daily and social activities, questioning what activities and how often they do in stroke patients. While the first 10 items ask individuals to estimate the frequency of household chores such as preparing meals and washing clothes in the last 3 months, the next 5 items ask them to indicate the frequency of social activities such as travel and gardening in the last six months. Response scores range from 0 (never) to 3 (at least 1 per week). The total scoring range is between 0 (no participation) and 45 (frequent participation).
Stroke-specific quality of life | through study completion, an average of 6 month
  The Stroke-Specific Quality of Life Scale consists of 49 items and 12 domains to assess the quality of life of individuals diagnosed with stroke. These areas are; mobility (6 items), energy (3 items), upper extremity function (5 items), work production (3 items), temperament (5 items), self-care (5 items), social role (5 items), family role ( 3 items), vision (3 items), language (5 items), thinking (3 items) and personality traits (3 items). The items were graded with a Likert-type scoring ranging from 1 to 5. Rating was made as 1. Strongly agree, 2. Partially agree, 3. Undecided, 4. Partially disagree, 5. Strongly disagree. A high scale score indicates a high quality of life, and a low scale score indicates a low quality of life.
Exercise benefits and barriers | through study completion, an average of 6 month
  The Benefits / Barriers of Exercise Scale consists of 24 items, 2 open-ended questions and six sub-dimensions. While 12 of the 24 items of the scale consist of statements about the benefits of exercise, the other 12 are made up of statements that prevent exercise. Negative items are coded in reverse. The scale is evaluated with a 4-point Likert scale. It is scored as 4 (Strongly Agree), 3 (Agree), 2 (Disagree), and 1 (Strongly Disagree). The scale is evaluated over the total score (min=24, max= 96). Higher scores indicate a perception of greater exercise benefits and less exercise barriers.
Exercise behaviour | through study completion, an average of 6 month
  Behavioral Regulations in Exercise Scale-2 consists of 19 items and five subscales. These are: external regulation, introjective regulation, identification regulation, internal regulation and amotivation subscales. The Behavioral Regulations in Exercise Scale-2 is a 5-point Likert-type scale with a score between 0-4, consisting of "not at all true", "sometimes true" and "definitely true". Increasing and decreasing scores according to the sub-scales express positive and negative behavioral thoughts.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only researchers in the study will have access to individual data.